CLINICAL TRIAL: NCT03891186
Title: A Randomized Controlled Trial to Evaluate the Efficacy of Metacognitive Training for Schizophrenia Applied by Mental Health Nurses: Study Protocol
Brief Title: Efficacy of Metacognitive Training for Schizophrenia - a Study Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Rovira i Virgili (Other)
Collaborators: Center for Health Technology and Services Research (Other)
Responsible Party: Principal Investigator, Carme Ferré Grau, Professor, University Rovira i Virgili
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2019MCT.PT
Record Dates: First submitted 2019-02-05; First posted 2019-03-26 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Schizophrenia
Keywords: schizophrenia; metacognitive training; insight; positive symptoms; functioning
MeSH Terms: conditions — Schizophrenia | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Metacognitive Training For Schizophrenia
Who Masked: Investigator, Outcomes Assessor
Masking Description: Eligible participants will be recruited by the investigators in collaboration with the multidisciplinary team of each institution. A baseline assessment will be carried out and the instruments will be applied after informed consent by participants. Participants will be randomly allocated to either Metacognitive Training (MCT) (experimental group). The control group will not participate in the MCT program. In both groups will be maintained the TAU. The variables for whom the participants are stratified are educational level, duration of mental disorder and type of treatment. All participants will be re-assessed at the end of the program and three months later. The program will be applied during four weeks (two session per week).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Participants will be randomly allocated to either Metacognitive Training (MCT) (experimental group). In both groups will be maintained the "treatment as usual" (TAU).
  Interventions: Behavioral: Metacognitive Training in Schizophrenia (MCT); Other: Treatment As Usual (TAU)
- Control Group (Active Comparator): The control group will not participate in the MCT program. In both groups will be maintained the TAU.
  Interventions: Other: Treatment As Usual (TAU)

INTERVENTIONS:
Behavioral: Metacognitive Training in Schizophrenia (MCT) — MCT is a group program with eight modules referring to common cognitive and biases in solving problems in schizophrenia. The following topics of MCT are: attribution blaming and taking credit (module 1), jumping to conclusions (modules 2 and 7), changing beliefs (module 3), deficits in theory of mind and social cognition (modules 4 and 6), overconfidence in (memory) errors (module 5) and depression and low self-esteem (module 8). Each session lasts 45 to 60 minutes and follows a protocol defined in the manual "Metacognitive Training for Psychosis (MCT)" that is currently available in 35 languages (available in www.uke.de/mkt).
  Arms: Experimental Group
Other: Treatment As Usual (TAU) — In both groups will be maintained the TAU.

SUMMARY:
Metacognitive training (MCT) for schizophrenia has been used in several countries, but its efficacy remains unclear. MCT is a program group that consists of changing the cognitive infrastructure of delusions.

This study aims to evaluate the efficacy of the Portuguese version of the metacognitive training programme and its effects on psychotic symptoms, insight to the disorder and functionality

DETAILED DESCRIPTION:
A randomized controlled trial that will be realized in six psychiatric institutions of Portugal. Pilot study will be carried out initially. The sample will be constituted by individuals diagnosed with schizophrenia (experimental group (n=30) and control group (n=30). The evaluation instruments will be utilized are PSYRATS, BCIS, PSP and WHODAS 2.0 applied to both groups in three different moments. In experimental group the eight MCT modules will be applied over four weeks.

The objective is to compare the outcomes associated with "treatment-as-usual" and the benefits of implementing the Metacognitive Training for Schizophrenia.

The hypothesis to be validated in this trial are:

* the schizophrenic patients who integrate the experimental group and participate in the MCT program will reduce the severity of psychotic symptoms and will present a better insight to disease and a better functioning on the final of the program than the control group;
* in participants that participating in the MCT program, the psychotic symptoms decrease at the end of the program and in the follow up (three months later) and the awareness for the disease and functioning improves.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 65 years;
* diagnosis of schizophrenia evaluated by Psychiatrist Assistant;
* that didn't have any changes in neuroleptics medication four months before program.

Exclusion Criteria:

* substance dependence;
* very severe psychotic symptoms that impedes understanding the objectives of the sessions;
* had changes in neuroleptics medication four months before program.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2020-04-04 (Actual); Study Completion 2020-04-04 (Actual)

PRIMARY OUTCOMES:
Psychotic Symptom Rating Scales (PSYRATS) - moment 1 | PSYRATS will be applied a week before the first session of Metacognitive Training.
  This instrument is a structured interview that assesses the detailed measurement of delusions and hallucinations. The PSYRATS have 17 items and two subscales: one subscale assesses delusions (6 items) and the other subscale assess hallucinations (11 items). Each item has a classification of five points (0-4). The total score is the sum of all points. It is was developed by Haddock, McCarron, Tarrier and Faragher in 1999 (validated for the Portuguese population by Telles-Correia et al in 2017).
Psychotic Symptom Rating Scales (PSYRATS) - moment 2 | PSYRATS will be applied up to 1 week after eight session, to both groups.
  This instrument is a structured interview that assesses the detailed measurement of delusions and hallucinations. The PSYRATS have 17 items and two subscales: one subscale assesses delusions (6 items) and the other subscale assess hallucinations (11 items). Each item has a classification of five points (0-4). The total score is the sum of all points. It is was developed by Haddock, McCarron, Tarrier and Faragher in 1999 (validated for the Portuguese population by Telles-Correia et al in 2017).
Psychotic Symptom Rating Scales (PSYRATS) - moment 3 | This instrument will be reapplied to follow up evaluation, up to 3 months after the final program, in both groups.
  This instrument is a structured interview that assesses the detailed measurement of delusions and hallucinations. The PSYRATS have 17 items and two subscales: one subscale assesses delusions (6 items) and the other subscale assess hallucinations (11 items). Each item has a classification of five points (0-4). The total score is the sum of all points. It is was developed by Haddock, McCarron, Tarrier and Faragher in 1999 (validated for the Portuguese population by Telles-Correia et al in 2017).
Beck Cognitive Insight Scale (BCIS) - moment 1 | BCIS will be applied a week before the first session of Metacognitive Training
  This scale has 15 items and it is a self-response questionnaire that was developed by Beck, Baruch, Balter, Steer, & Warman in 2004 and evaluated the consciousness of the illness. The BCIS is comprised of two subscales: self-reflectiveness and self-certainty. The total score for each scale is the sum of the item scores that comprise it (see below). The BCIS composite index is calculated as self-reflectiveness minus self-certainty. Poorer cognitive insight is indexed by lower scores on the self-reflectiveness subscale, higher self-certainty scores, and lower BCIS composite index scores.
  Step 1. Score every item on the BCIS from "0" to "3" according to the following rule:
  * "Do Not Agree at All" = 0
  * "Agree Slightly" = 1
  * "Agree a Lot" = 2
  * "Agree Completely" = 3 (in process of validation to Portuguese population by investigators of this study)
Beck Cognitive Insight Scale (BCIS) - moment 2 | BCIS will be applied up to 1 week after eight session of the MCT, to both groups
  This scale has 15 items and it is a self-response questionnaire that was developed by Beck, Baruch, Balter, Steer, & Warman in 2004 and evaluated the consciousness of the illness. The BCIS is comprised of two subscales: self-reflectiveness and self-certainty. The total score for each scale is the sum of the item scores that comprise it (see below). The BCIS composite index is calculated as self-reflectiveness minus self-certainty. Poorer cognitive insight is indexed by lower scores on the self-reflectiveness subscale, higher self-certainty scores, and lower BCIS composite index scores.
  Step 1. Score every item on the BCIS from "0" to "3" according to the following rule:
  * "Do Not Agree at All" = 0
  * "Agree Slightly" = 1
  * "Agree a Lot" = 2
  * "Agree Completely" = 3 (in process of validation to Portuguese population by investigators of this study)
Beck Cognitive Insight Scale (BCIS) - moment 3 | This instrument will be reapplied to follow up evaluation, up to 3 months after the final program in both groups.
  This scale has 15 items and it is a self-response questionnaire that was developed by Beck, Baruch, Balter, Steer, & Warman in 2004 and evaluated the consciousness of the illness. The BCIS is comprised of two subscales: self-reflectiveness and self-certainty. The total score for each scale is the sum of the item scores that comprise it (see below). The BCIS composite index is calculated as self-reflectiveness minus self-certainty. Poorer cognitive insight is indexed by lower scores on the self-reflectiveness subscale, higher self-certainty scores, and lower BCIS composite index scores.
  Step 1. Score every item on the BCIS from "0" to "3" according to the following rule:
  * "Do Not Agree at All" = 0
  * "Agree Slightly" = 1
  * "Agree a Lot" = 2
  * "Agree Completely" = 3 (in process of validation to Portuguese population by investigators of this study)
World Health Disability Assessment Schedule (WHODAS 2.0) - moment 1 | WHODAS 2.0 will be applied a week before the first session of Metacognitive Training
  This instrument evaluated the functionality levels and was developed by WHO. It has 12 items and it is a self-response questionnaire (validated for the Portuguese population by Moreira, Alvarelhão, Silva, Costa and Queirós in 2015).
World Health Disability Assessment Schedule (WHODAS 2.0) - moment 2 | WHODAS 2.0 will be applied up to 1 week after eight session of the MCT, to both groups
  This instrument evaluated the functionality levels and was developed by WHO. It has 12 items and it is a self-response questionnaire (validated for the Portuguese population by Moreira, Alvarelhão, Silva, Costa and Queirós in 2015).
World Health Disability Assessment Schedule (WHODAS 2.0) - moment 3 | This instrument will be reapplied to follow up evaluation, up to 3 months after the final program in both groups.
  This instrument evaluated the functionality levels and was developed by WHO. It has 12 items and it is a self-response questionnaire (validated for the Portuguese population by Moreira, Alvarelhão, Silva, Costa and Queirós in 2015).
Personal and Social Performance Scale (PSP) - moment 1 | PSP will be applied a week before the first session of Metacognitive Training
  this scale was developed by Morosini, Magliano, Brambilla, Ugolini and Pioli in 2000 and it assesses patients' social functioning with four main areas: socially useful activities, personal and social relationships, self-care and disturbing and aggressive behaviours (validated for the Portuguese population by Brissos et al., 2012).
Personal and Social Performance Scale (PSP) - moment 2 | PSP will be applied up to 1 week after eight session of the MCT, to both groups
  this scale was developed by Morosini, Magliano, Brambilla, Ugolini and Pioli in 2000 and it assesses patients' social functioning with four main areas: socially useful activities, personal and social relationships, self-care and disturbing and aggressive behaviours (validated for the Portuguese population by Brissos et al., 2012).
Personal and Social Performance Scale (PSP) - moment 3 | This instrument will be reapplied to follow up evaluation, up to 3 months after the final program in both groups.
  this scale was developed by Morosini, Magliano, Brambilla, Ugolini and Pioli in 2000 and it assesses patients' social functioning with four main areas: socially useful activities, personal and social relationships, self-care and disturbing and aggressive behaviours (validated for the Portuguese population by Brissos et al., 2012).

OTHER OUTCOMES:
Sociodemographic and clinical data | Sociodemographic and clinical data will be applied a week before the first session of Metacognitive Training on both groups.
  Age, gender (male (1) or female (2)), marital status (single (1), married (2), divorced (3), widower (4)), cohabitation (institution (1), alone (2), parents (3), mother or father (4), son (5), sibling (6), other family (7), other non-family (8)), educational level (illiterate (1), primary education (2), 6th grade (3), 9th grade (4), Secondary education (5), Bachelor (6), Master degree (7), PhD (8)), professional/employment status (employee (1), unemployed (2), disability (3), retired (4), medical leave (5)), duration of mental disorder (< 1 year (1), 1 to 2 years (2), 2 to 5 years (3), 5 to 10 years (4), 10 to 20 years (5), > 20 years ago (6)), number of Psychiatric hospitalizations (only once (1), 2 to 5 times (2), 6 to 10 times (3), more than 10 times (4)) and substance use (tobacco (1), alcohol (2), other drugs(3)). This data will be collected a week before be beginning program to all participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Lara Manuela Guedes de Pinho, Portalegre, Portugal

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] de Pinho LMG, Sequeira CADC, Sampaio FMC, Rocha NB, Ozaslan Z, Ferre-Grau C. Assessing the efficacy and feasibility of providing metacognitive training for patients with schizophrenia by mental health nurses: A randomized controlled trial. J Adv Nurs. 2021 Feb;77(2):999-1012. doi: 10.1111/jan.14627. Epub 2020 Nov 22. PMID 33222210